CLINICAL TRIAL: NCT06043245
Title: Prognostic Factors and Predictors of Diabetes Remission in Hypoabsorptive Bariatric Surgery Techniques. Randomized Comparative Study Between Duodenal Switch, Single-Anastomosis Duodenal Switch (SADI-S) and Mini-Gastric Bypass
Brief Title: Diabetes Remission and Hypoabsorptive Bariatric Surgery
Acronym: DIABAR-3
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Nuria Vilarrasa, Principal Investigator, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR015/23
Record Dates: First submitted 2023-06-11; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Severe Obesity; Diabetes Mellitus, Type 2; Bariatric Surgery Candidate
Keywords: Diabetes remission; hypoabsortive bariatric surgery; Incretin hormones; Gut microbiota
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus, Type 2 | interventions — Anastomosis, Surgical

STUDY DESIGN:
Intervention Model Description: Three parallel groups (patients with severe obesity and Type 2 Diabetes) assigned 1:1:1 to undergo duodenal switch (DS), Single anastomosis duodeno-ileal (SADI-S) or Minigastric bypass (MGB).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Duodenal switch (Active Comparator): The restrictive portion of the surgery involves removing approximately 70% of the stomach (along the greater curvature) and most of the duodenum. The malabsorptive portion of the surgery reroutes a lengthy portion of the small intestine, creating two separate pathways and one common channel.The common channel is 200 cm and 100m the alimentary limb.
  Interventions: Procedure: Duodenal Switch
- SADI-S (Active Comparator): Creation of a sleeve gastrectomy (SG) and a duodenal-ileal anastomosis with preservation of the pylorus, jejunal exclusion and a total common-alimentary limb, originally measuring 200 cm and later standardized to 300 cm to reduce the risk of nutritional deficiencies.
  Interventions: Procedure: SADI-S
- Minigastric bypass (Active Comparator): Creation of a gastric pouch similar to Sleeve gastrectomy and the small bowel is run to 200 cm distal to Treitz' ligament and then anastomosed antecolic end-to-side to the gastric pouch.
  Interventions: Procedure: Minigastric Bypass

INTERVENTIONS:
Procedure: Duodenal Switch — Classic Duodenal Switch
  Arms: Duodenal switch
Procedure: SADI-S — SADI-S with a 300cm common channel
  Other Names: Single- Anastomosis Duodenal Switch
  Arms: SADI-S
Procedure: Minigastric Bypass — Classic minigastric bypass
  Other Names: Single anastomosis or Omega loop gastric bypass
  Arms: Minigastric bypass

SUMMARY:
Bariatric surgery is the most effective treatment to achieve type 2 Diabetes Mellitus (DM) remission in patients with severe obesity. However, there is little evidence of the effectiveness and pathophysiological mechanisms involved in metabolic improvement after hypoabsortive tecniques such as duodenal switch (DS), single anastomosis duodenal switch (SADI-S) or minigastric bypass (MGB). We have designed a randomized study to compare type 2 diabetes remission after the 3 bariatric procedures in patients with severe obesity (BMI > 45kg/m2) and to study the implication of gastrointestinal hormones, bile acids and gut microbiota in metabolic improvement in each procedure.

DETAILED DESCRIPTION:
Patients fulfilling inclusion criteria will be randomly assigned 1:1:1 to undergo DS, SADI-S or MGB. Allocation of patients will be assigned by simple randomization with stratification according to baseline levels of HbA1c (greater or lower/ equal to 7 %).

Protocol 0. Screening visit: All participants will be required to sign the informed consent, according to the regulations of the Committee of the center. Clinical, analytical, and general physical examination data will be collected and it will be checked the fulfillment of inclusion criteria.

1. Visit 1 (1 week after screening visit): Anthropometrical data will be collected, and general biochemical analytics including HbA1c, lipid profile and nutritional parameters and vitamins will be performed. Also a standard meal test (SMT) will be done with determination of GLP-1, PYY, GIP , and ghrelin, insulin, glucose and succinate concentrations before and during the SMT. A complete body composition study including DEXA, BIA and cardiac resonance to determine epicardia fat will be performed. Feces samples will be collected to determine gut microbiota. Quality of live questionnaire will be provided.
2. Visit2 (1 month after surgery): Glycaemia diaries will be checked. Anthropometrical, general biochemical analysis with determination of HbA1c, lipid profile and nutritional parameters and vitamins will be done. SMT will be performed with determination of GLP-1, PYY, GIP, ghrelin, insulin, glucose. A determination of bile acids will be done before starting the meal test. feces samples will be collected to determine gut microbiota.
3. Visit 3 (3 months after surgery): Glycaemia diaries will be checked. Anthropometrical, general biochemical analysis with determination of HbA1c, lipid profile and nutritional parameters and vitamins will be done.
4. Visit 4 (12 months after surgery): The same determinations of visit 1 will be performed 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* BMI>45 kg/m2
* T2D on treatment with hypoglycemic agents alone, insulin or both.

Exclusion Criteria:

* Type 1 diabetes
* Positivity for GAD auto-antibodies
* Secondary forms of diabetes
* Acute metabolic complications in the last 6 months
* Severe liver disease
* Renal dysfunction
* Patients under anticoagulant treatment
* Previous bariatric surgery
* Congenital or acquired abnormalities of the digestive tract
* Pregnancy
* Nursing or desired pregnancy in the 12 months following inclusion
* Corticoid use by oral or intravenous route for more than 14 consecutive days in the last three months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Type 2 Diabetes (T2D) remission. | 12 months
  Number of participants achieving T2D remission (HbA1c <6.5% without anti-diabetic treatment) in each arm group one year after surgery.

SECONDARY OUTCOMES:
Weight loss | 12 months
  Percentage of total weight loss from baseline to 12 months after surgery in the three arm groups
Entero-endocrine hormone GLP-1 | 12 months
  Changes in plasma concentrations of gut hormone GLP-1 from baseline to 12 months after surgery in the three arm groups
Entero-endocrine hormone PYY | 12 months
  Changes in plasma concentrations of gut hormone PYY from baseline to 12 months after surgery in the three arm groups
Entero-endocrine hormone GIP | 12 months
  Changes in plasma concentrations of gut hormone PYY from baseline to 12 months after surgery in the three arm groups
Entero-endocrine hormone Ghrelin | 12 months
  Changes in plasma concentrations of gut hormone Ghrelin from baseline to 12 months after surgery in the three arm groups
Bile salts | 12 months
  Changes in plasma concentrations of primary and secondary bile salts from baseline to 12 months after surgery in the three arm groups
Intestinal microbiome | 12 months
  Changes in the ratio of Firmicutes and bacteroidetes species from baseline to 12 months after surgery in the three arm groups
Epicardial fat | 12 months
  Changes in epicardial fat from baseline to 12 months after surgery measured in mm2 in the three arm groups

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Vilarrasa García, PhD, MD, Principal Investigator — Medical doctor at Hospital Universitari de Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finno P, Osorio J, Garcia-Ruiz-de-Gordejuela A, Casajoana A, Sorribas M, Admella V, Serrano M, Marchesini JB, Ramos AC, Pujol-Gebelli J. Single Versus Double-Anastomosis Duodenal Switch: Single-Site Comparative Cohort Study in 440 Consecutive Patients. Obes Surg. 2020 Sep;30(9):3309-3316. doi: 10.1007/s11695-020-04566-5. PMID 32240495
- [Result] Gebelli JP, Lazzara C, de Gordejuela AGR, Nora M, Pereira AM, Sanchez-Pernaute A, Osorio J, Sobrino L, Garcia AJT. Duodenal Switch vs. Single-Anastomosis Duodenal Switch (SADI-S) for the Treatment of Grade IV Obesity: 5-Year Outcomes of a Multicenter Prospective Cohort Comparative Study. Obes Surg. 2022 Dec;32(12):3839-3846. doi: 10.1007/s11695-022-06317-0. Epub 2022 Oct 25. PMID 36282430